CLINICAL TRIAL: NCT05425576
Title: Phase 2 Trial of TGF-β Inhibition (OT-101) With Anti-PD-1 (Pembrolizumab) in Patients With Malignant Pleural Mesothelioma (MPM) Failing to Achieve or Maintain Response to Checkpoint Inhibition
Brief Title: OT-101 in Combination With Pembrolizumab in Subjects With Malignant Pleural Mesothelioma Failing to Respond to Checkpoint Inhibition
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oncotelic Inc. (Industry)
Responsible Party: Sponsor
Organization: Mateon Therapeutics (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OT-01-M201
Record Dates: First submitted 2022-06-09; First posted 2022-06-21 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Malignant Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug OT-101 plus pembrolizumab (Experimental): OT-101 will be administered at a RP2D dose/m2/day for 4 days continuously and 10 days off every two weeks via a portable infusion pump.
  Pembrolizumab will be administered with the standard regimen of 400 mg intravenously (IV) every six weeks.
  Interventions: Drug: OT-101

INTERVENTIONS:
Drug: OT-101 — OT-101 in combination of pembrolizumab
  Other Names: Pembrolizumab

SUMMARY:
This is a study of OT-101, a TGF-b2 inhibitor in combination of pembrolizumab in patients with malignant pleural mesothelioma. Both efficacy assessment, and safety and tolerability of various dose of OT-101 in combination of pembrolizumab are evaluated.

DETAILED DESCRIPTION:
This is a phase 2, open label, non-randomized, single arm Simon's two stage study in subjects with malignant pleural mesothelioma failing to achieve or maintain response to checkpoint inhibition. Before the efficacy assessment portion, the study will first embark a run-in dose-escalation phase to evaluate safety and tolerability of various dose of OT-101 in combination of pembrolizumab, and to determine a recommended Phase 2 dose (RP2D) of 4 days continuous I.V. infusion for every two weeks regimen. Subjects received the RP2D in the run-in dose-escalation phase will be part of the first stage of the Simon's two-stage design for effectiveness evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have progressed on treatment with an anti-PD-1 or anti-PD-L1 mAb or anti-CTLA-4 mAb administered either as monotherapy or in combination with other therapies including platinum-based chemotherapy. PD-1 treatment progression is defined by meeting all of the following criteria:

   a. Has demonstrated disease progression after anti-PD-1 or anti-PD-L1 or anti-CTLA-4 mAb as defined by the investigator.
2. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of Malignant Pleural Mesothelioma will be enrolled in this study.
3. Male participants: A male participant must agree to use contraception as detailed in Appendix 4 of this protocol during the treatment period and for at least 90 days, corresponding to time needed to eliminate any study treatment(s) (e.g. 5 terminal half-lives for pembrolizumab) plus an additional 90 days (a spermatogenesis cycle) for study treatments with evidence of genotoxicity at any dose after the last dose of study treatment and refrain from donating sperm during this period.
4. Female participants: A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) OR
   2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 90 days/weeks corresponding to time needed to eliminate any study treatment(s) plus 30 days (a menstruation cycle) for study treatments with risk of genotoxicity after the last dose of study treatment.
5. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
6. Have measurable disease by Revised mRECIST
7. Provide a baseline biopsy prior to the start of therapy. Archival biopsy is acceptable.
8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
9. Have adequate organ function. Specimens must be collected within 10 days prior to the start of study intervention.

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to agent administration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior systemic anti-cancer therapy including investigational agents within 28 days prior to study therapy.
3. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
4. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
5. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug. The following are exceptions to this criterion:

   * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
   * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
   * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
6. Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years.
7. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 10 days prior to first dose of study intervention.
8. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
10. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
11. Has an active infection requiring systemic therapy.
12. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
16. Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Determination of ORR for the combination of OT-101 and pembrolizumab in subjects | approximately 24 months
  modified RECIST (mRECIST; v1.1)

SECONDARY OUTCOMES:
PFS, DOR and 6-month and 12-month Overall Survival (OS) will be estimated in all subjects in the ITT population. | approximately 18 months
  Progression-free Survival (PFS), defined as the time from date of first dose of study drug to date of documented PD based on modified RECIST v1.1.
  Duration of Response (DOR), defined as the time from date of first documented response (CR or PR) to date of documented progressive disease (PD), based on modified RECIST v1.1.
  Overall Survival (OS), defined as the time from the date of first dose of study drug to the date of death.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States